CLINICAL TRIAL: NCT04190667
Title: A Study on the Homologous Recombination Deficiency Status in Chinese Population With Epithelial Ovarian Cancer
Brief Title: Homologous Recombination Deficiency Status in Epithelial Ovarian Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Lei Li (Other)
Responsible Party: Sponsor-Investigator, Lei Li, Professor, Peking Union Medical College Hospital
Organization: Peking Union Medical College Hospital (Other)
Other Study IDs: EOC-HRD
Record Dates: First submitted 2019-12-04; First posted 2019-12-09 (Actual); Last update posted 2019-12-10 (Actual); Status verified 2019-12

CONDITIONS: Epithelial Ovarian Cancer; Chinese; Homologous Recombination Deficiency; BRCA1 Mutation; BRCA2 Mutation; Prognosis
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial | interventions — Genetic Profile

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Samples from the patients' peripheral blood and tumor tissues.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Genomic testing — A multi-panel testing of 36 genes would be given for these patients in their peripheral blood and tumor tissues. These 36 genes include: BRCA1, BRCA2, ABRAXAS1(FAM175A）, ATM, ATR, BAP1, BARD1, BRIP1, C11ORF30（EMSY）, CDK12, CHEK1, CHEK2, FANCA, FANCC, FANCD2, FANCI, FANCL, MRE11A, NBN, PALB2, PPP2R2A, PTEN, RAD50, RAD51B, RAD51C, RAD51D, RAD54B, RAD54, MLH1, MSH2, MSH6, PMS2, EPCAM, STK11, TP53, CDH1. The study would select 150 patients with pathogenic or likely pathogenic mutations in BRCA1/2 and 150 patients without these mutations to further explore the HRD status.

SUMMARY:
The homologous recombination deficiency (HRD) status in Chinese population with epithelial ovarian cancer (EOC) is little known. This study would recruit 1300 Chinese EOC patients. A multi-panel testing of 36 genes would be given for these patients in their peripheral blood and tumor tissues. These 36 genes include: BRCA1, BRCA2, ABRAXAS1(FAM175A）, ATM, ATR, BAP1, BARD1, BRIP1, C11ORF30（EMSY）, CDK12, CHEK1, CHEK2, FANCA, FANCC, FANCD2, FANCI, FANCL, MRE11A, NBN, PALB2, PPP2R2A, PTEN, RAD50, RAD51B, RAD51C, RAD51D, RAD54B, RAD54, MLH1, MSH2, MSH6, PMS2, EPCAM, STK11, TP53, CDH1. The study would select 150 patients with pathogenic or likely pathogenic mutations in BRCA1/2 and 150 patients without these mutations to further explore the HRD status. The HRD model is based on the loss of heterozygosity (LOH), telomere allele imbalance (TAI) and large-scale state transitions (LST). The mutated genes, HRD score model and their relationship with the prognosis, would provide a full description of for the Chinese EOC patients.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older
* Pathological confirmation of epithelial ovarian cancer
* With available tumor tissues
* Given consents to participate the study

Exclusion Criteria:

* Not meeting all of the inclusion criteria

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chinese population with confirmed diagnosis of epithelial ovarian cancer
Sampling Method: Non-Probability Sample
Enrollment: 1300 (Estimated)
Dates: Start 2019-12-07 (Actual); Primary Completion 2021-12-07 (Estimated); Study Completion 2022-12-07 (Estimated)

PRIMARY OUTCOMES:
Frequency of targeted genetic mutations | Two years
  Frequency of pathogenic or likely pathogenic mutations in a multi-panel genes
Homologous recombination deficiency (HRD) score | Two years
  The HRD score for individual patient is a scale describing her HRD status. The score model is calculated by the analysis for three types of important molecular mechanism: loss of heterozygosity (LOH), telomere allele imbalance (TAI) and large-scale state transitions (LST)

SECONDARY OUTCOMES:
Progression-free survival | Two years
  Progression-free survival in recruited patients
Overall survival | Two years
  Overall survival in recruited patients
Rate of sensitivity to platinum-based chemotherapy | Two years
  Sensitivity to platinum-based chemotherapy in recruited patients
Rate of sensitivity to poly-(ADP-ribose) polymerase inhibitors | Two years
  Sensitivity to poly-(ADP-ribose) polymerase inhibitors in recruited patients

CONTACTS AND LOCATIONS:
Overall Officials: Lei Li, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Lei Li, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided